CLINICAL TRIAL: NCT05964270
Title: The Impact of Telemonitoring on Correct Drug Use, Complications and Quality of Life Among Patients With Multiple Myeloma (MM)
Brief Title: Telemonitoring Among Patients With Multiple Myeloma
Acronym: ITUMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Job Eijsink, Principal Investigator, Isala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ITUMM
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
Keywords: Value-base health care; e-coach; adherence
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: A two-arm open-label parallel-group randomized controlled trial (RCT) will be conducted at a supra regional cancer center (referred to as 'het oncologisch centrum Isala'), which provides hematology services to a population with 0.5 million adherence and a population of 1 million referral, in the Northern-East region of The Netherlands.
Who Masked: Care Provider
Masking Description: pill count
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Active Comparator): participants of the intervention group (IG) will get a login for the e-coach MM, and access to eight modules: medication, outpatient visit preparation, periodic assessment, messaging service, alerts, information, ad hoc complaint, personal care plan. IG participants information is collected on a web platform that automatically invites enrolled patients. The e-coach MM is available 24/7.
  Interventions: Device: e-coach multipel myeloma (MM)
- Control group (CG) (No Intervention): Participants in the CG (control group) will only get a login for a 'dummy version' without the modules, besides the periodic assessments (questionnaires), at the same time as the IG

INTERVENTIONS:
Device: e-coach multipel myeloma (MM) — In this study we developed a multimodal patient-centered MM e-coach between September 2019 and June 2020. The content of the intervention consist of eight modules and was tested in a pilot study between June 2020 and August 2020 (F-ITUMM) 22. The e-coach is digitally managed, following three phases of the tiers of VBHC as presented in Figure 1. The tiers are classified in health status, process of recovery and sustainability of health 30. Furthermore, all medication information plus current dose and frequency per unit time are integrated in the e-coach. Reminders are sent if a session or a medication unit time is exceeded. Feasibility was tested for patients as well as healthcare professionals. The F-ITUMM trial concluded that the MM e-coach has the potential to support both recently diagnosed MM patients and healthcare professionals during MM treatment, and is a promising application to improve adherence .
  Arms: Intervention group (IG)

SUMMARY:
A two-arm open-label parallel-group randomized controlled trial will be conducted to compare the telemonitoring (MM e-coach) with standard MM care. This study aimed to recruit 150 patients with recently diagnosed multiple myeloma (RDMM), starting first or second line of treatment. Blinded primary outcome is adherence by pill count after start of treatment at 1-3 months. Secondary outcomes are patient reported outcomes: Groninger frailty index (GFI), quality of life (EQ-5D-5L, EORTC-QLQ-C30), shared decision making (SDM-Q-9), self-reported adherence (MARS-5), single item questions, patient experiences (PREMs), adverse events, overall survival (OS) and progression free survival (PFS). Patient reported outcomes were developed and integrated in the e-coach MM to regularly measure digitized outcomes of MM patients from time of RDMM until 12 months post-diagnosis. Online measurements will be performed at baseline (0), 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a participant (patient) must meet all of the -following criteria:

* signed informed consent
* >18 years
* recently diagnosed MM patients with first-line or second-line treatment
* able to complete patient-reported outcome measures and experiences
* have minimal digital skills to check if they are able to interact with an e-coach
* can read and understand Dutch.

Participants who meet any of the following criteria will be excluded from participation in this study

* psychiatric illness requiring secondary-care intervention
* too ill to engage with the intervention in the opinion of the clinical care team
* no perspective of >12 months survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
blinded primary outcome by pill count | over a time periode of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Job Eijsink, PharmD, Principal Investigator — Isala klinieken department clinical pharmacy
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Eijsink JFH, Geerts PAF, Kamminga K, Edens MA, Boersma C, Postma MJ, Maring JG, Ter Horst PGJ. The impact of telemonitoring on correct drug use, complications and quality of life among patients with multiple myeloma (ITUMM): A study protocol for an open-label, parallel-group, randomized controlled trial. PLoS One. 2024 Aug 26;19(8):e0307177. doi: 10.1371/journal.pone.0307177. eCollection 2024. PMID 39186588